CLINICAL TRIAL: NCT04818476
Title: Outcomes of Endoscopically Resected High-risk Mucosal Adenocarcinoma and Low- and High-risk Submucosal Adenocarcinoma Arising in Barrett's Esophagus: an International Multicenter Retrospective Cohort Study
Brief Title: Outcomes of Endoscopically Resected High-risk Mucosal and Low- and High-risk Submucosal Adenocarcinoma Arising in Barrett's Esophagus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, prof. dr. J.J.G.H.M. Bergman, Professor of Gastrointestinal Endoscopy, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: x
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Barrett Esophagus; Adenocarcinoma Esophagus; Submucosal Esophageal Adenocarcinoma; High-risk Mucosal Esophageal Adenocarcinoma
Keywords: Barrett Esophagus; Submucosal esophageal adenocarcinoma; Endoscopic treatment; Endoscopic follow-up; High-risk mucosal esophageal adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HR-T1a: Patients who weretreated by radical endoscopic resection for a high-risk mucosal EAC (HR-T1a N0M0)
  Interventions: Procedure: diagnostic endoscopic resection
- LR-T1b: Patients who were treated by radical endoscopic resection for a low-risk submucosal EAC (LR-T1b N0M0)
  Interventions: Procedure: diagnostic endoscopic resection
- HR-T1b: Patients who were treated by radical endoscopic resection for a high-risk submucosal EAC (HR-T1b N0M0)
  Interventions: Procedure: diagnostic endoscopic resection

INTERVENTIONS:
Procedure: diagnostic endoscopic resection — diagnostic endoscopic resection

SUMMARY:
The purpose of this study is to assess lymph node metastasis rate, distant metastasis rate, disease-specific mortality, and overall mortality in patients with Barrett's related T1b and high risk T1a esophageal adenocarcinoma (EAC) who underwent a diagnostic endoscopic resection.

DETAILED DESCRIPTION:
The incidence of esophageal adenocarcinoma (EAC) has increased six-fold over the last three decades, making it the most rapidly rising cancer in the Western world. The main histologic risk factor for development of EAC is the presence of Barrett's esophagus (BE). BE can develop from non-dysplastic BE, to low (LGD) and high grade dysplasia (HGD) and, eventually, EAC.

The past two decades minimally invasive endoscopic resection (ER) has replaced surgical esophagectomy as first-choice therapy for the treatment of early neoplastic lesions in Barrett's esophagus. ER provides adequate tissue specimens, allowing for accurate histopathological staging of a lesion, by assessment of invasion depth, differentiation grade, presence of lympho-vascular invasion (LVI), and radicality of the resection. Endoscopic resection thus similarly fulfils a diagnostic and therapeutic role in the management of Barrett's neoplasia.

However, ER offers local treatment and does not include lymph node dissection as is still standard of care during esophagectomy. Therefore, the choice to perform endoscopic follow-up after a radical ER of an early EAC, or to refer a patient for additional surgery, is guided by the assumed risk of lymph node metastasis (LNM).

Data from previous studies show that the risk of LNM is only 1% in patients with low risk mucosal EAC after endoscopic treatment (i.e., infiltration depth limited to the mucosa, G1-G2, without LVI), and <2% in low risk submucosal EAC (i.e., infiltration depth <500μm, good to moderate differentiation grade (G1-G2), without LVI). In high risk submucosal EAC (i.e., infiltration depth ≥500 μm, and/or G3-G4, and/or LVI), the LNM risk is estimated to be much higher (16-44%). Nevertheless, these numbers are mainly based on old surgical series.

Current data is limited in terms of small and heterogeneous patient cohorts, and data for patients with high risk T1a EAC is not available at all. Therefore, we would like to conduct an international multicenter retrospective cohort study in >10 centers to evaluate the safety and efficacy of endoscopic treatment and follow-up of patients with high risk mucosal and submucosal EAC. Our main focus will be the presence of lymph node metastasis and EAC related death.

Aim of this registration study is to collect data of the above-mentioned group of patients and thereby assess lymph node metastasis rate, disease-specific mortality, and overall mortality.

This study will be conducted according to the principles of the Declaration of Helsinki and in accordance with the Medical Research Involving Human Subjects Act (WMO), the Medical Treatment Contracts Act (WGBO) and the Dutch Personal Data Protection Act (WBP). The investigators will perform the study in accordance with this protocol and will make sure that participants do not object to using their data. Collection, recording, and reporting of data will be accurate and will ensure the privacy, health, and welfare of research subjects during and after the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, all ages
2. Endoscopic resection of a histologically proven high risk T1a, low risk T1b EAC, or high risk T1b EAC
3. Between 1/1/2008 and 1/1/2019
4. Endoscopic resection and endoscopic FU (or other treatment after ER) have taken place in the participating center
5. No written or oral refusal to use subject's data

Exclusion Criterium:

Objection against participation in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent a diagnostic ER for Barrett's related HR T1a or T1b EAC in one of the participating centers, from 1/1/2008 up to the moment of data collection.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
lymph node metastasis rate | 10 years
  Confirmed by cytology and/or histology by performing FNA during EUS or biopsies
distant metastasis rate | 10 years
  Primary tumor of distant metastasis should be histopathologically evalueted by taking biopsies.
disease-specific mortality | 10 years
  Disease specific mortality is decribed as mortality directly linked to the esophageal adenocarcinoma (i.e., metastasized EAC, metastasized disease with a simultaneously primary cancer present and it cannot be ruled out (based on histology) that the metastases are related to the other primary cancer, death due to complications of the endoscopic procedure, death due to complications after surgery or CRT, no clear cause of death in patients who have metastases or untreated local recurrence). If patients are diagnosed with distant metastases, and subsequently die of a non-tumor related cause, patients will still be documented as tumor-related death. Will be measured in number of patients and percentages. Survival analysis using Kaplan Meier will be performed.
overall mortality | 10 years
  Overall mortality of study population (tumor-related + non-tumor-related deaths). Measured in numbers and percentages, survival analysis (KM).

CONTACTS AND LOCATIONS:
Overall Officials: R.E. Pouw, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (16):
- Westmead hospital, Sydney, Australia
- UZ Gasthuisberg, Leuven, Belgium
- CHU Nantes, Nantes, France
- Germany (4):
  - Universitätsklinikum Augsburg, Augsburg
  - EVK Duesseldorf, Düsseldorf
  - MRI TUM, Münich
  - Barmherzige Brüder Regensburg, Regensburg
- Netherlands (7):
  - Amsterdam UMC, location VUmc, Amsterdam
  - Catharina Hospital, Eindhoven
  - University Medical Center Groningen, Groningen
  - St. Antonius Hospital, Nieuwegein
  - Erasmus MC - University Medical Center, Rotterdam
  - Haga Medical Center, The Hague
  - Isala Clinics, Zwolle
- Hirslanden private hospital group, Zurich, Switzerland
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No